CLINICAL TRIAL: NCT01856270
Title: Amitriptyline to Prevent Headache After Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jeanne Hoffman, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001333
Record Dates: First submitted 2013-05-10; First posted 2013-05-17 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Brain Injuries; Post-Traumatic Headache
Keywords: Traumatic brain injury; Post-traumatic headache; Drug therapy
MeSH Terms: conditions — Brain Injuries; Post-Traumatic Headache; Brain Injuries, Traumatic | interventions — Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amitriptyline Immediate (Experimental): The Amitriptyline Immediate group will begin study drug immediately after enrollment. Immediate Drug participants will be started on one 10 mg capsule each evening. The dosage will be adjusted upwards to 25 mg daily for Week 2 to a maximum of 50 mg daily by Week 3.
  Interventions: Drug: Amitriptyline
- Amitriptyline Delayed (Experimental): The Amitriptyline Delayed group will start the study drug at the Day 30 visit on one 10 mg capsule each evening. The dosage will be adjusted upwards to 25 mg daily for Week 2 to a maximum of 50 mg daily by Week 3.
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline — Participants with headache will be enrolled within the first 12 weeks after injury and will be randomly assigned to 2 groups (see Table 1 for summary of protocol). Group 1 will be assessed within 3 months of injury (baseline, Day 0) (when they will receive their initial ramp-up dosage containers; see Table 2 for dosing), Day 30 and Day 60 (to monitor compliance and distribute study drug), and for final outcome on Day 90. Group 2 will be assessed within 3 months of injury (baseline, Day 0) but will not receive medication until their Day 30 visit. Those in group 2 who report headache at Day 30 will receive their initial dosage container and will then be reassessed at Day 60 (to monitor compliance and distribute study drug) and Day 90 (final outcome).
  Other Names: Elavil

SUMMARY:
The investigators propose to conduct a 2-arm, open-label pilot study to determine if early treatment with amitriptyline will decrease the frequency and severity of headaches after mild traumatic brain injury (TBI). Amitriptyline is a tricyclic antidepressant that is commonly available and inexpensive. It is used as a first-line drug for primary headache prevention in a very low dose range of 10-50 mg.

* Specific Aim 1 is to conduct a 2-arm open-label study to examine the effect of preventive treatment with amitriptyline on the frequency and severity of headache after mild TBI.
* Specific Aim 2 is to collect data needed for design of a Phase 3 study, including an estimate of effect size, headache variability, and desirable drug treatment start date.
* Specific Aim 3 is to examine the feasibility of using headache diaries with individuals with mild TBI.
* Specific Aim 4 is to establish the safety and tolerability of amitriptyline for the prevention of headache after mild TBI.

The investigators hypothesize that early preventive treatment with amitriptyline will avert the development of chronic post-traumatic headache (PTH) as compared to rates of headache from a recent natural history study on PTH after mild TBI.

The investigators propose to enroll inpatient subjects from a Level I trauma center as well as from outpatient clinics and from the general community with a diagnosis of mild TBI. Subjects will be screened for current headache. After baseline assessment, 72 subjects with current headache will be randomized to one of 2 groups. Group 1 will immediately begin amitriptyline and or Group 2 will be followed and begin amitriptyline at Day 30. All subjects will be asked to complete a daily headache diary beginning on Day 1 of the study. A detailed medical history and headache survey will be completed. Subjects will have a scheduled stepped increase in the drug dosage every week for 3 weeks to the maximum study dosage of 50 mg. Weekly telephone calls will monitor for adverse events and compliance with the drug and headache diary. Clinic visits will occur at 30, 60 and 90 days. The 30 day clinic visit will include cognitive testing to assess for differences between groups and initiation of drug treatment for Group 2. Both 30 and 60 day visits will include review of headache diary, potential adverse effects, and pill counts. The 90 day visit will be for outcome assessment. In addition, the headache survey will be repeated by telephone at Day 180.

DETAILED DESCRIPTION:
Research Hypothesis and Aims: The ultimate aim of this research is to determine whether early treatment using amitriptyline can prevent the development of chronic headache after TBI. This proposal is for preliminary work that will give some indication of the effect of amitriptyline and provide information needed to design a definitive study of the efficacy of amitriptyline for the prevention of chronic post-traumatic headache.

Specific Aim 1 is to conduct a two-arm open-label study to examine the effect of preventive treatment with amitriptyline on the frequency and severity of headache after mild TBI compared to that seen in our observational study on the natural history of headache after mild TBI.

Specific Aim 2 is to collect data needed for design of a Phase III study, including an estimate of effect size, the variability in the number of headache days in those with mild TBI, and determining a desirable initiation date for preventive treatment (e.g., week 1 or month 1 after injury).

Specific Aim 3 is to examine the feasibility of headache diary use in individuals with mild TBI.

Specific Aim 4 is to establish the safety and tolerability of amitriptyline for the prevention of headache after mild TBI.

Hypothesis: Preventive treatment of early headaches with amitriptyline after mild TBI results in decreased prevalence of recurrent headache (percent of participants having at least 1 headache/week) and severe headaches (percent of participants having headaches with an average pain of 5 or higher) at three months as compared to the frequency and severity of headache in those followed in the natural history study who received usual care.

Data Collection and Measures: Data collection will occur at enrollment, at each clinic visit, and at Day 180. An examiner blinded to group assignment will administer all measures at Clinic Visit 1 as cognition will be compared between groups at that time point; other assessment points will be unblinded.

Primary Outcome Measure: Frequency and severity of headaches at 90 days after study initiation.

Secondary Measures: Secondary measures are the Brief Pain Inventory, Analog Pain Scale, Pain Sites, Headache Impact Test-6 (HIT-6), Insomnia Severity Index (ISI), Patient Health Questionnaire-9 (PHQ-9), General Anxiety Disorder - 7 Item Scale (GAD-7), Alcohol Use Disorders Identification Test-Consumption (AUDIT-C), Rivermead Post-Concussion Symptom Questionnaire (RPQ), EuroQol, Health Survey Short Form-12® (SF-12), and Satisfaction with Life Scale. Caffeine use and drug use questions will be asked that will model the AUDIT questions. Additional measures will be obtained at baseline to characterize injury type and severity, medication use, and accompanying disorders.

Headache Diary: The subject will be asked to fill out a headache diary each day during the study to rate the frequency and severity of headache as well as some simple headache characterization.

Enrollment and Randomization: Informed consent will be obtained from the participant as approved by the Human Subjects Division of the University of Washington. Subjects will be randomized into one of two groups (Group 1: early start vs. Group 2: delayed start) using a computerized blocked randomization, stratified on headache severity (average severity of <4 vs. >5).

Medication administration and dosing adjustments: The study drug, amitriptyline, will be dispensed in medication containers clearly marked with the dosage and instructions to take at bedtime daily (separate containers for 10 mg, 25 mg, and 50 mg). Once randomized, Group 1 participants will be started on one 10 mg capsule each evening. The dosage will be adjusted upwards to 25 mg daily for Week 2 to a maximum of 50 mg daily by Week 3. Group 2 participants will be assessed on Clinic Visit 1 (Day 30) for current headache. If the participant has continued to have headaches (new or worse than pre-injury), he/she will have the same ramp-up schedule when the study drug is started at Day 30. Those in group 2 who do not have headaches at day 30 will be followed by phone and with headache diaries throughout the study including outcomes. If the perceived side effects of the study drug are intolerable at any time during the study, subjects will be asked to decrease the dosage to half a pill until a new prescription arrives. If side effects remain intolerable after 3 days on the lower dose, that subject will be discontinued from the study drug but followed in the study. Regardless of dose, the schedule for visits and testing will continue. Participants will be allowed to use rescue medications as needed for headache.

Compliance: Each dosage will be in a separate pill container and clearly marked. Compliance will be assessed during the weekly telephone follow-up calls and at the follow-up clinic visits. Pill counts will be performed at each visit. Adequate compliance will be considered 80% medication consumption.

Schedule of Visits: Baseline Hospital Visit. Measures administered will include an interim medical history form (diagnoses, current medications), headache survey, pain measures, HIT-6, PHQ-9, ISI, RPQ, and SF-12. After completion of baseline assessments, the research assistant will instruct the participant in the use of a daily headache diary. The research assistant will distribute the labeled study drug to each Group 1 participant and will instruct on use. Participants will be given a schedule for increasing the dose weekly. Subjects will be asked to keep their pill containers to turn in at the next clinic visit.

Telephone Follow-Up Calls 1-9 (between clinic visits). The research assistant will contact the participant weekly (Telephone Follow-Up Calls 1, 2, 3) after enrollment to check on completion of headache diary and to confirm frequency and severity of headaches during the preceding week, study drug use, and use of rescue medications. In the case of adverse effects which are bothersome to the patient (e.g., mild sedation, dry mouth, constipation), the dosage will be decreased by one dosage level or by ½ pill per day.

Clinic Visit 1 (Day 30). For all participants on this visit, vital signs will be obtained. Drug containers will be collected from Group 1 and headache diaries will be collected from all subjects. Measures administered on this visit will include an interim medical history form (new diagnoses, changes in medications), headache survey, pain measures, HIT-6, PHQ-9, ISI, RPQ,and SF-12. Neuropsychological tests will be given on this visit only. For Group 1, if the dosage was decreased secondary to minor adverse events in the interim, one of the study physicians will meet with the participant to decide whether to maintain a lower dose or have a second trial of returning to a higher dose of the study drug. The second month's supply of study drug will be dispensed at this visit. For Group 2 participants with headache, medications for the first month of treatment will be distributed along with a ramp-up schedule.

Clinic Visit 2 (Day 60). Vital signs will be obtained. Drug containers and headache diaries will be collected from all subjects. Measures administered on this visit will include an interim medical history form (new diagnoses, changes in medications), headache survey, pain measures, HIT-6, PHQ-9, ISI, RPQ, and SF-12. If the dosage was decreased secondary to minor adverse events in the interim, one of the study physicians will meet with the participant to decide whether to maintain a lower dose or have a second trial of returning to a higher dose of the study drug. The final month's supply of study drug will be dispensed at this visit.

Clinic Visit 3 (Day 90). This will be the final visit for the subjects. Vital signs will be obtained. Drug containers and headache diaries will be collected from all subjects. Measures administered on this visit will include an interim medical history form (new diagnoses, changes in medications), headache survey, pain measures, HIT-6, PHQ-9, ISI, RPQ,and SF-12.

Telephone Follow-Up Call 10. The research assistant will call the subject at Day 180 to administer the headache survey (which includes the HIT-6) and record current medications only.

Subject Withdrawal: Subjects may be discontinued from the study drug on their request or if the subject experiences an adverse effect sufficient to warrant withdrawal from the study drug, In the case of discontinuation, the reason for withdrawal will be recorded and the subject will be asked to continue to monitor their headaches with use of the headache diary.

Data Analysis Study Sample Size and Rationale: In a recent observational study, the investigators observed that of people with new or worse headaches at baseline assessment after mild TBI, 35% had 1 or more headaches per week at 3 months and a similar fraction had average headache pain severity of 6 or more on a 0 (no pain) to 10 (worst pain imaginable) scale. The study's two end points are: 1) reduction in the percent of people with baseline headaches that has one or more headaches per week at 3 months; and 2) the reduction in the percent of people with baseline headaches that experience headache severity of 6 or more on a scale from 0 to 10 at 3 months. It will be necessary for 65 cases to be followed to 3 months in order to have 80% power to reject the null hypothesis of a 35% headache rate if amitriptyline taken as a preventive yields 21% of subjects having 1 or more headaches per week (a 40% reduction in the percentage of people with frequent headaches at 3 months). Similar numbers are needed to confirm a like reduction in the percent of participants with severe headaches (average pain of 6 or greater). These are based on a 1-sided significance level of 0.05. Allowing for up to 10% attrition (7 subjects), the investigators will recruit and randomize 72 participants. Based on the previous natural history study, the investigators expect about 104 cases per year to have new or worse headaches at baseline assessment. The investigators expect 60% to meet the eligibility criteria and 60% of those to consent to participate, yielding 37 cases per year to randomize.

Aim 1. The primary intent-to-treat analysis will determine the proportion of participants with frequent (1 or more headaches per week) or severe (with average pain of 6 or higher) headaches combining both arms at 3 months. Each of these proportions will be compared to the rate of each recorded in our observational study using a normal approximation to the binomial (one-sided chi-squared test). In the previous observational study, the investigators observed 35% with at least 1 headache per week and 36% with headaches having average pain of at least 6 on a scale from 0 to 10. A one-sided significance level of 0.05 will be used. The investigators will also examine evidence for any differential benefit for amitriptyline started at baseline or 1 month to help decide which to use for the Phase III trial if this pilot suggests that is worthwhile.

Aim 2. Descriptive statistics will be used (means, standard deviations, proportions) to help in the planning of the Phase II trial.

Aim 3 (feasibility of use of a headache diary). This will be addressed by examining the number of participants who do not use their diary at all, have over 10% missing data, or who report different values on the phone calls than is shown in the diary. Different modes of completing the diary (paper, smart phone or web application) will be studied to see if any are more user friendly for this population.

Aim 4. Descriptive statistics will be used to summarize the occurrence of adverse events. The investigators will estimate the impact of amitriptyline on cognition by comparing the neuropsychological performance at 1 month of those started on the drug at baseline to those who start drug after the 1-month assessment. The mean difference on each test will be calculated with a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Acute mild TBI (Glasgow Coma Scale of 13-15 on emergency department evaluation, any period of loss of consciousness (LOC) < than 30 minutes, alteration of consciousness or post-traumatic amnesia (not to exceed 24 hours)
* Ability to give consent
* Ages 18-60
* Access to a telephone
* Current headache (new headache or headache worse than prior to injury)

Exclusion Criteria:

* Does not speak English
* Diagnosed seizure disorder
* Myocardial infarction in prior 6 months
* Cardiac arrhythmia requiring medication treatment
* Prolonged Q-T interval on electrocardiogram
* Psychosis
* Intoxication on hospital admission sufficient enough to cloud the diagnosis of mild TBI
* Incarceration or homelessness
* Allergy to amitriptyline
* Current treatment with amitriptyline or other tricyclic antidepressant
* Currently taking any medication not recommended for use with amitriptyline due to the potential for Q-T interval prolongation. Examples of this include: Class I, I-A or II antiarrhythmics, TCA's, MAOI's, selected fluoroquinolones (gatifloxacin, moxifloxacin), selected antipsychotic medications (haloperidol, risperidone, quetiapine), selected antiretroviral medications, cisapride, chloroquine, chlorpromazine, prochlorperazine, promethazine, citalopram, fluoxetine, erythromycin, methadone
* History of glaucoma
* History of prostate disease or current urinary retention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Hoffman, PhD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Amitriptyline Immediate: The Immediate group will begin study drug immediately after enrollment. Immediate Drug participants will be started on one 10 mg capsule each evening. The dosage will be adjusted upwards to 25 mg daily for Week 2 to a maximum of 50 mg daily by Week 3.
  Amitriptyline: Participants with headache will be enrolled within the first 12 weeks after injury and will be randomly assigned to 2 groups. Group 1 will be assessed within 3 months of injury (baseline, Day 0) (when receiving initial ramp-up dosage containers), Day 30 and 60 (to monitor compliance and distribute study drug), and for final outcome on Day 90. Group 2 will be assessed within 3 months of injury (baseline, Day 0) but will not receive medication until Day 30 visit. Those in group 2 who report headache at Day 30 will receive their initial dosage container and will then be reassessed at Day 60 (to monitor compliance/distribute study drug) and Day 90 (final outcome).
- Amitriptyline Delayed: The Delayed group will start the study drug at the Day 30 visit on one 10 mg capsule each evening. The dosage will be adjusted upwards to 25 mg daily for Week 2 to a maximum of 50 mg daily by Week 3.
  Amitriptyline: Participants with headache will be enrolled within the first 12 weeks after injury and will be randomly assigned to 2 groups. Group 1 will be assessed within 3 months of injury (baseline, Day 0) (when they will receive their initial ramp-up dosage containers), Day 30 and Day 60 (to monitor compliance and distribute study drug), and for final outcome on Day 90. Group 2 will be assessed within 3 months of injury (baseline, Day 0) but will not receive medication until their Day 30 visit. Those in group 2 who report headache at Day 30 will receive their initial dosage container and will then be reassessed at Day 60 (to monitor compliance and distribute study drug) and Day 90 (final outcome).
Period: Overall Study
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed
Started | 24 | 26
Completed (Completed the 180 day assessment) | 13 | 14
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Amitriptyline Immediate: The Immediate group will begin study drug immediately after enrollment. Immediate Drug participants will be started on one 10 mg capsule each evening. The dosage will be adjusted upwards to 25 mg daily for Week 2 to a maximum of 50 mg daily by Week 3.
  Amitriptyline: Participants with headache will be enrolled within the first 12 weeks post injury and will be randomly assigned to 2 groups. Group 1 will be assessed within 3 months of injury (baseline, Day 0) (when they will receive their initial ramp-up dosage containers), Day 30 and 60 (to monitor compliance/distribute study drug), and for final outcome on Day 90. Group 2 will be assessed within 3 months of injury (baseline, Day 0) but will not receive medication until Day 30 visit. Those in group 2 who report headache at Day 30 will receive initial dosage container and reassessed at Day 60 (to monitor compliance and distribute study drug) and Day 90 (final outcome).
- Amitriptyline Delayed: The Delayed group will start the study drug at the Day 30 visit on one 10 mg capsule each evening. The dosage will be adjusted upwards to 25 mg daily for Week 2 to a maximum of 50 mg daily by Week 3.
  Amitriptyline: Participants with headache will be enrolled within the first 12 weeks post injury and will be randomly assigned to 2 groups. Group 1 will be assessed within 3 months of injury (baseline, Day 0) (when they will receive their initial ramp-up dosage containers), Day 30 and 60 (to monitor compliance/distribute study drug), and for final outcome on Day 90. Group 2 will be assessed within 3 months of injury (baseline, Day 0) but will not receive medication until their Day 30 visit. Those in group 2 who report headache at Day 30 will receive initial dosage container and then reassessed at Day 60 (to monitor compliance and distribute study drug) and Day 90 (final outcome).
- Total: Total of all reporting groups
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (11.7) | 34.6 (12.7) | 35.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 11 | 17 | 28
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Headaches
Description: Number of subjects reporting an average of at least one headache per week
Time Frame: 90 days
Population: The two arms are combined for this analysis to answer the question of frequency of headache at the 3 month outcome data point and only difference between arms was related to onset time of medication which was not expected to result in significant change in headache frequency, but only potentially in cognitive status.
Measure: Count of Participants; unit: Participants
Groups:
- Amitriptyline Sample: Individuals enrolled into the study and who have completed headache diaries through 3 months post injury.
Arm/Group | Amitriptyline Sample
Number analyzed (Participants) | 43
Participants | 10
Statistical Analysis 1: Comparison: Amitriptyline Sample; A positive difference of proportions would indicate an improvement in the Amitriptyline sample, while a negative difference would indicate a worsening; Test type: Superiority — The data from this study was compared with the data from the Natural History of Headache after Mild TBI which was previously published (Lucas, Hoffman, Bell, Dikmen. (2014), A prospective study of prevalence and characterization of headache following mild traumatic brain injury. Cephalalgia (34) 93-102); p = .101, Fisher Exact — A priori significance threshold α=.05; Difference of proportions = 0.114, 95% CI 1-sided [lower limit -0.017] — Confidence interval estimation method from Wallenstein (1997). 71 of 205 participants (at 3 Mo post) in the Natural History study endorsed having a headache more than once per week

2. Primary Outcome: Severity of Headache
Description: Number of subjects with headache reporting an average pain of at least 6 on a 0-10 scale with 0=no pain and 10=worst pain.
Time Frame: 90 days
Population: The two arms are combined for this analysis to answer the question of severity of headache at the 3 month outcome data point and only difference between arms was related to onset time of medication which was not expected to result in significant change in headache frequency, but only potentially in cognitive status.
Measure: Count of Participants; unit: Participants
Groups:
- Amitriptyline Study: Individuals enrolled into the current study.
Arm/Group | Amitriptyline Study
Number analyzed (Participants) | 38
Participants | 7
Statistical Analysis 1: Comparison: Amitriptyline Study; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .017, Fisher Exact — A priori significance threshold α=.05; Difference of proportions = .194, 95% CI 1-sided [lower limit .057] — Confidence interval estimation method from Wallenstein (1997). 56 of 148 participants (at 3 mo post) in the Natural History study reported pain >=6

3. Secondary Outcome: Number of Participants With Adverse Events Possibly Related to Study Medication
Description: The number and types of treatment related adverse events will be monitored on a weekly basis and will be divided by severity if differing.
Time Frame: Day 1 through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed
Number analyzed (Participants) | 24 | 26
Participants
  Number wth any events | 5 | 3
  # with Possible, probable or definite rel to tx | 4 | 1
  # with tx related moderate/severe events | 0 | 0
Statistical Analysis 1: Comparison: Amitriptyline Immediate vs Amitriptyline Delayed; Test type: Superiority; p = .456, Fisher Exact — A priori significance threshold α=.05; Difference of proportions = .093, 95% CI 2-sided [-.106 to .286] — Estimate is the effect observed in the Immediate group (i.e. Immediate - Delayed). Confidence interval estimation method from Wallenstein (1997)

4. Secondary Outcome: Rey Auditory Verbal Learning Test (Total)
Description: The Rey Auditory Verbal Learning Test will be administered at 30 days to detect potential changes in cognitive function due to study drug. Scoring is based on the total number of words recalled from a list of 15 across 5 trials (max score of 75) with higher score indicating better learning.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: words recalled
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed
Number analyzed (Participants) | 12 | 11
words recalled | 26.3 (4.7) | 27.1 (5.0)
Statistical Analysis 1: Comparison: Amitriptyline Immediate vs Amitriptyline Delayed; Test type: Superiority; p = .684, t-test, 2 sided — A priori significance threshold α=.05; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-5.1 to 3.4] — Estimate is the effect observed in the Immediate group (i.e. Immediate - Delayed)

5. Secondary Outcome: Rey Auditory Verbal Learning Test (Short)
Description: The Rey Auditory Verbal Learning Test will be administered at 30 days to detect potential changes in cognitive function due to study drug. Scoring is based on the total number of words recalled from the original list of 15 after a new list of 15 is given (used as distraction). Higher scores indicate better short-term memory.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: words recalled
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed
Number analyzed (Participants) | 12 | 11
words recalled | 10.3 (1.8) | 9.4 (2.5)
Statistical Analysis 1: Comparison: Amitriptyline Immediate vs Amitriptyline Delayed; Test type: Superiority; p = .306, t-test, 2 sided — A priori significance threshold α=.05; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-1.0 to 2.9] — Estimate is the effect observed in the Immediate group (i.e. Immediate - Delayed)

6. Secondary Outcome: Rey Auditory Verbal Learning Test (Long)
Description: The Rey Auditory Verbal Learning Test will be administered at 30 days to detect potential changes in cognitive function due to study drug. Scoring is based on the total number of words recalled from the original list of 15 after a 30 minute time delay. Higher scores indicate better long-term memory.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: words recalled
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed
Number analyzed (Participants) | 10 | 11
words recalled | 13.6 (1.3) | 13.3 (1.4)
Statistical Analysis 1: Comparison: Amitriptyline Immediate vs Amitriptyline Delayed; Test type: Superiority; p = .583, t-test, 2 sided — A priori significance threshold α=.05; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.9 to 1.6] — Estimate is the effect observed in the Immediate group (i.e. Immediate - Delayed)

7. Secondary Outcome: Trail Making Test (A)
Description: Trail Making Test will be given at 30 days to detect any impact of study drug on cognition. This is a test of visual attention and is scored by the number of seconds it takes to complete the task of making a trail through letters.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed
Number analyzed (Participants) | 12 | 11
seconds | 28.7 (9.0) | 26.3 (5.3)
Statistical Analysis 1: Comparison: Amitriptyline Immediate vs Amitriptyline Delayed; Test type: Superiority; p = .444, t-test, 2 sided — A priori significance threshold α=.05; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-4.0 to 8.8] — Estimate is the effect observed in the Immediate group (i.e. Immediate - Delayed)

8. Secondary Outcome: Trail Making Test (B)
Description: Trail Making Test will be given at 30 days to detect any impact of study drug on cognition. This is a test of visual attention and task switching and is scored by number of seconds it takes to complete the task (switching from letters to numbers in order).
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed
Number analyzed (Participants) | 11 | 11
seconds | 87.5 (34.9) | 60.3 (21.3)
Statistical Analysis 1: Comparison: Amitriptyline Immediate vs Amitriptyline Delayed; Test type: Superiority; p = .041, t-test, 2 sided — A priori significance threshold α=.05; Mean Difference (Final Values) = 27.3, 95% CI 2-sided [1.2 to 53.3] — Estimate is the effect observed in the Immediate group (i.e. Immediate - Delayed)

9. Secondary Outcome: Wechsler Adult Intelligence Scale (WAIS) IV Digit Symbol
Description: The WAIS IV Digit Symbol test will be given to detect any effect of study drug on cognition. This test assesses processing speed and new learning and requires an individual to substitute the relevant digit for a symbol and are given a time limit. The total number of correct digits are summed and converted to a scaled score (range 1-20 with 10 being at the 50th percentile) with higher scores indicating better performance.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: standard score
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed
Number analyzed (Participants) | 12 | 12
standard score | 7.5 (2.5) | 9.3 (2.3)
Statistical Analysis 1: Comparison: Amitriptyline Immediate vs Amitriptyline Delayed; Test type: Superiority; p = .089, t-test, 2 sided — A priori significance threshold α=.05; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.8 to 0.3] — Estimate is the effect observed in the Immediate group (i.e. Immediate - Delayed)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of medication usage at baseline, then at day 30, day 60, and at day 90 when medication was discontinued.
Groups:
- Amitriptyline Immediate: The Immediate group will begin study drug immediately after enrollment. Immediate Drug participants will be started on one 10 mg capsule each evening. The dosage will be adjusted upwards to 25 mg daily for Week 2 to a maximum of 50 mg daily by Week 3.
- Amitriptyline Delayed: The Delayed group will start the study drug at the Day 30 visit on one 10 mg capsule each evening to assess whether there is any cognitive impact of the medication (comparing to those who started immediately after enrollment. The dosage will be adjusted upwards to 25 mg daily for Week 2 to a maximum of 50 mg daily by Week 3.
Arm/Group | Amitriptyline Immediate | Amitriptyline Delayed
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 5/24 | 3/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amitriptyline Immediate (N=24) | Amitriptyline Delayed (N=26)
Dry Mouth (Gastrointestinal disorders) | 3 (4) | 0 (0)
Groggy (Nervous system disorders) | 0 (0) | 1 (1)
Increased QTc (Cardiac disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (2) | 1 (1)
decreased libido (Renal and urinary disorders) | 1 (1) | 0 (0)
possible metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
sleep difficulties (Nervous system disorders) | 1 (1) | 0 (0)
respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a prevention study recruiting from hospital inpatients or from the ED with a diagnosis of mild TBI. We were unable to recruit an adequate number of subjects and had difficult follow up. Of those recruited, we followed only 54%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No